CLINICAL TRIAL: NCT02395705
Title: A Phase III, Multicenter Randomized Controlled Study of Neo-adjuvant Chemotherapy Paclitaxel + Cisplatin Versus Surgery Alone for Stage IIA-IIIB Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant Chemotherapy Versus Surgery Alone for Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Peking University Cancer Hospital & Institute (Other); Hunan Province Tumor Hospital (Other); Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yin Li, Vice-President, Director of thoracic surgery department, Henan Cancer Hospital, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Henan CH
Record Dates: First submitted 2015-02-26; First posted 2015-03-24 (Estimated); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Esophageal Neoplasm
MeSH Terms: conditions — Esophageal Neoplasms | interventions — TP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neo-adjuvant chemotherapy group (Experimental): Neo-adjuvant chemotherapy(cisplatin and paclitaxel):
  1. Paclitaxel, 175mg/m2, d1, Cisplatin, 25mg/m2, d2-d4, 3 week, 2 cycles.
  2. Paclitaxel, 87.5mg/m2, d1,d8, Cisplatin, 25mg/m2, d2-d4, 3 week, 2 cycles.
  3. Paclitaxel, 175mg/m2, d1, Cisplatin, 75mg/m2, d1, 3 week, 2 cycles.
  Surgery:
  2-3weeks after Neo-adjuvant chemotherapy
  1. Surgeons: the operation shall be performed by senior thoracic surgeons. Try to achieve the consistency of operation quality.
  2. Operation: the thoracic esophagectomy must be through right thoracic cavity. (open and minimally invasive McKeown or Ivor Lewis). Total two-field lymphadenectomy (right and left recurrent laryngeal nerve lymph nodes must be included).
  Interventions: Drug: cisplatin and paclitaxel
- Surgery alone group (No Intervention): Surgery:
  2-3weeks after Neo-adjuvant chemotherapy
  1. Surgeons: the operation shall be performed by senior thoracic surgeons. Try to achieve the consistency of operation quality.
  2. Operation: the thoracic esophagectomy must be through right thoracic cavity. (open and minimally invasive McKeown or Ivor Lewis). Total two-field lymphadenectomy (right and left recurrent laryngeal nerve lymph nodes must be included).

INTERVENTIONS:
Drug: cisplatin and paclitaxel — 1. Paclitaxel, 175mg/m2, d1, Cisplatin, 25mg/m2, d2-d4, 3 week, 2 cycles.
  2. Paclitaxel, 87.5mg/m2, d1,d8, Cisplatin, 25mg/m2, d2-d4, 3 week, 2 cycles.
  3. Paclitaxel, 175mg/m2, d1, Cisplatin, 75mg/m2, d1, 3 week, 2 cycles.
  Other Names: TP
  Arms: Neo-adjuvant chemotherapy group

SUMMARY:
The effect of neo-adjuvant chemotherapy on survival of patients with thoracic esophageal squamous cell carcinomas remains the most controversial part of neo-adjuvant therapy for esophageal carcinomas. One of our objectives is to evaluate whether the neo-adjuvant therapy with cisplatin and paclitaxel followed by right thoracic approach esophagectomy with total 2-field lymph node dissection improves the overall survival of thoracic esophageal cancer patients.

DETAILED DESCRIPTION:
The effect of Neo-adjuvant chemotherapy on survival of patients with thoracic esophageal squamous cell carcinomas remains the most controversial part of Neo-adjuvant therapy for esophageal carcinomas. Therefore, the optimal management of resectable esophageal squamous cell carcinomas differs widely among different areas based on local randomized controlled trials.

The neo-adjuvant chemotherapy might be a good strategy if sufficient local control is achieved by surgical treatment. This study defined the detail of surgery procedure and the region of lymphadenectomy and adopted cisplatin and paclitaxel as neoadjuvant chemotherapy regimens. We try to evaluate the efficacy and safety of this neo-adjuvant strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of squamous cell thoracic esophageal carcinoma of Stage IIA to IIIB, (7th Union for International Cancer Control, UICC-TNM).
2. Patients must not have received any prior anticancer therapy of esophageal carcinoma.
3. Age ranges from 18 to 75 years.
4. Without operative contraindication.
5. Absolute white blood cells count ≥4.0×109/L, neutrophil ≥1.5×109/L, platelets ≥100.0×109/L, hemoglobin ≥90g/L, and normal functions of liver and kidney, total bilirubin（TBIL）≤1.5N, aspartate aminotransferase (AST)≤2.5N, alanine aminotransferase(ALT)≤2.5N, prothrombin time(PT)≤1.5N, and activated partial thromboplastin time(APTT) is in normal range, endogenous creatinine clearance rate(CRE)≤1.5N.
6. Patients must not have diagnosed with other cancer and must not received any prior anticancer therapy except prostatic cancer with more than 5 years disease-free survival(DFS).
7. expected R0 resection.
8. ECOG 0～2.
9. Signed informed consent document on file. 10.No metastatic lymph node in cervical by color doppler sonography.

Exclusion Criteria:

1. Multiple primary cancer.
2. The subject cannot understand and sign the informed consent form(ICF).
3. Patients with concomitant hemorrhagic disease.
4. Any un expected reason for patients can't get operation.
5. Inability to use gastric conduit after esophagectomy because of a prior surgery.
6. Pregnant or breast feeding.
7. Patients are diagnosed or suspected to be allergic to cisplatin or Paclitaxel.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | 5 years

SECONDARY OUTCOMES:
Overall survival rate | 1 years and 3 years
Disease free survival | 5 years
assessment in perioperation-Removal rate (R0 resection rate) | perioperative period
  The R0 resection rate of two groups
assessment in perioperation-Rate of Operative Complication | perioperative period
  Complication rate after operation before discharge
assessment in perioperation-Mortality of perioperation | perioperative period
  Mortality of perioperation 20 days before operation and 30 days after operation
assessment in perioperation-Days of Hospitalization | perioperative period
  Days of Hospitalization after operation
assessment in perioperation-Thoracic Drainage | perioperative period
  Thoracic Drainage days
assessment in perioperation-Quantity of bleeding | perioperative period
  blood lose during operation
assessment in perioperation-Time of operation | perioperative period
  the time from open thoracic cavity to the closure of the thoracic cavity
Quality of life | 1 years
  ECOG, KPS, NRS-2002, EORTC QLQ-ST018, EORTC QLQ-C30
efficacy of neo-adjuvant chemotherapy--response rate | 1-4 days before operation
  Criteria:Response Evaluation Criteria in Solid Tumors，RECIST. Pathologic Complete Response Rate. Pathologic Response Rate.
toxicities of neo-adjuvant chemotherapy | from chemotherapy to perioperative period
  According to National Cancer Institute Common Terminology Criteria for Adverse Event,Version 3.0(CTC AE3.0). The complete rate of protocol
prognostic factors | 5 years
  prognostic factors for overall survival of both groups
predictive factors | 2 years
  predictive factors for the efficiency of neo-adjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Yin Li, MD.&PhD., Principal Investigator — The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital
Locations (9):
- China (9):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-sen Uniersity Cancer Center, Guangzhou, Guangdong
  - Anyang cancer hospital, Anyang, Henan
  - Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan
  - Hunan Province Tumor Hospital, Changsha, Hunan
  - Fudan Universitay Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality